CLINICAL TRIAL: NCT04883294
Title: Validation of the Diagnostic Accuracy of the Electronic Nose in the Detection of Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL76036.068.21
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Thyroid Neoplasm
Keywords: Electronic Nose; Thyroid Neoplasm; Volatile Organic Compounds; Thyroid Cancer; Thyroid Nodule; Diagnosis
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Histology and Post-operative thyroid specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Group: A disease group including patients older than 18 years old with any kind of histopathologically proven malignancy of the thyroid gland (including Papillary thyroid cancer (PTC), Follicular thyroid cancer (FTC), Medullary thyroid cancer (MTC), and Anaplastic thyroid cancer);
  Interventions: Diagnostic Test: Electronic Nose
- Control: A control group including patients older than 18 years old with any kind of histopathologically proven benign thyroid gland disease (including adenoma, hyperplasia).
  Interventions: Diagnostic Test: Electronic Nose

INTERVENTIONS:
Diagnostic Test: Electronic Nose — All participants breathed through the Aeonose for five minutes. This device contains metal-oxide sensors that change in conductivity upon reaction with VOCs in exhaled breath. These conductivity changes are input data for machine-learning and used for pattern recognition. A nose clip was placed on the nose of each participant to avoid entry of non-filtered air in the device. Before measuring, the Aeonose was flushed with room air, guided through a carbon filter as well. Failed breath tests were excluded from analysis; the reason for failure was documented.
  Other Names: AeonoseTM

SUMMARY:
Patients with a suspected thyroid nodule face an invasive and patient unfriendly diagnostic work-up to determine the risk of malignancy. Typically, patients undergo ultrasound of the thyroid gland followed by fine-needle aspiration cytology (FNAC). FNAC has been considered as a gold standard diagnostic procedure in suspected thyroid nodules. Unfortunately, both the negative- and positive predictive value of FNAC is poor, often resulting in the need for a diagnostic hemithyroidectomy for definite diagnosis . Approximately 40-94% of the suspected thyroid nodules appear to be benign after resection and thus exposes patients to unnecessary surgery with unnecessary risks. Therefore, a quick, non-invasive assessment of the risk of malignancy of thyroid nodules is of paramount importance. Such a novel test could fasten the diagnostic process for patients with malignancies and reduce the amount of 'unnecessary' surgeries for benign conditions.

A promising development in cancer detection is based on volatile organic compounds (VOCs), gaseous degradation products of biochemical processes detectable in exhaled breath. During pathophysiological processes related to tumor growth, alterations in cell metabolism lead to a shift in the production of VOCs. The VOCs' patterns can be detected by the Aeonose™ through their reaction with the metal-oxide sensors in this device. A pilot study conducted at the Maastricht University Medical Center demonstrated that, by creating an artificial neural network (ANN) from the VOC patterns of numerous patients and their specific histopathological diagnosis, the Aeonose™ has a high diagnostic accuracy to discriminate benign from malignant thyroid nodules.

The purpose of this study is to validate the accuracy of the Aeonose™, to prevent unnecessary surgery and to investigate the use of the Aeonose™ as a surveillance tool in the postoperative follow-up of differentiated thyroid cancer.

We hypothesize that the high negative predictive value of the pilot study will be confirmed in the validation study and expect that implementation of the Aeonose™ in clinical practice will subsequently reduce the number of unnecessary surgeries below 10% for patients with Bethesda ≥ III nodules and may provide an important role in non-invasive detection of recurrent disease.

DETAILED DESCRIPTION:
Thyroid cancer is the most common endocrine cancer worldwide. In most developed countries, the incidence of thyroid cancer has rapidly increased in the last three decades In the Netherlands, 700 patients are diagnosed with thyroid cancer each year. The most common histological forms are the well-differentiated papillary and follicular cancer, comprising of 80-85% of all thyroid cancers

Patients often present themselves with a thyroid nodule, which can be benign or malignant. Current diagnostic work-up includes ultrasound of the neck, resulting in the Thyroid Imaging Reporting And Data System (TI-RADS). This risk-stratification system for thyroid nodules is based on ultrasound features. When indicated, fine-needle aspiration cytology (FNAC) is performed, resulting in the Bethesda classification to report the risk of malignancy. The FNAC has been considered as gold standard diagnostic procedure in suspected thyroid nodules . Unfortunately, both negative- and positive predictive value of FNAC is poor, often resulting in the need for a diagnostic hemithyroidectomy for definite diagnosis. 40-94% of the suspected thyroid nodules appear to be benign after resection. After surgical removal, patients with differentiated thyroid cancer sometimes receive adjuvant treatment with radioactive-iodine. Thereafter, patients face a long-term follow-up since recurrence of the disease may occur years after removal of the primary tumor. Based on risk stratification, serum thyroglobulin (Tg) levels are determined once or twice per year with or without additional imaging (e.g. thyroid ultrasound or total body scintigraphy). So, both diagnosis and follow-up of thyroid cancer are associated with invasive and unpleasant procedures for the patient.

After surgical removal, patients with differentiated thyroid cancer sometimes receive adjuvant treatment with radioactive-iodine. Thereafter, patients will be subjected to a long-term follow- up since recurrence of the disease may occur years after removal of the primary tumor. Based on risk stratification, serum thyroglobulin (Tg) levels are determined once or twice per year with or without additional imaging (e.g. thyroid ultrasound or total body scintigraphy). So, both diagnosis and follow-up of thyroid cancer are associated with invasive and unpleasant procedures for the patient.

A promising development in cancer detection is based on volatile organic compounds (VOCs), gaseous degradation products of biochemical processes detectable in exhaled breath. During pathophysiological processes related to tumor growth, alterations in cell metabolism lead to a shift in the production of VOCs. The VOCs' patterns can be detected by the Aeonose™ through their reaction to the metal-oxide sensors in this device. A pilot study conducted at the Maastricht University Medical Center+ demonstrated that, by creating an artificial neural network (ANN) from the VOC patterns of numerous patients and their specific histopathological diagnosis, the Aeonose™ has a high diagnostic accuracy to discriminate benign from malignant thyroid nodules.

The purpose of this study is to validate the accuracy of the Aeonose™, to prevent unnecessary surgery and to investigate the use of the Aeonose™ as a surveillance tool in the postoperative follow-up of differentiated thyroid cancer.

Aim

This study consists of three aims:

1. Confirm the results of the pilot study on the use of the Aeonose™ to distinguish benign from malignant thyroid nodules in a multicenter validation study.
2. Implement the use of the Aeonose™ in clinical practice, aiming to reduce unnecessary surgeries to <10%.
3. Investigate the use of the Aeonose™ to detect recurrent thyroid cancer in a patient friendly, non-invasive way compared to regular follow-up in a pilot study.

We plan to conduct an international prospective, observational multicenter study in twelve hospitals in the Netherlands, Belgium and Germany to validate the diagnostic performance of the Aeonose™ and to investigate its efficacy in the follow-up of differentiated thyroid cancer. First, a database of breathing patterns will be built to develop an ANN. An external validation study will be conducted using exhaled breath patterns of a total of 500 patients to address the first aim. Data from the validation study together with clinical parameters will be used to determine the necessity for a diagnostic hemithyroidectomy. The number of unnecessary surgeries will be evaluated. To address the third aim, a pilot study will be conducted. Patients with histologically proven differentiated thyroid cancer are asked to breathe in the Aeonose™ parallel to every regular follow-up moment. The Aeonose™ will be trained by the input of data of patients developing a recurrence or not to develop an ANN that can be used as a surveillance tool to detect recurrence non-invasively.

Before starting the validation study, the artificial neural network (ANN) that has been built in the pilot study will be expanded in the training study. The more patients included with a variety in breathing patterns (as a result of e.g. gender, age, smoking-status, food intake, medication use), the more stable and robust the model becomes. For this training study, a total of 200 patients with histopathological proven differentiated thyroid cancer is needed. Assuming that the prevalence of thyroid cancer among suspected thyroid nodules is 20%, a total of 1000 patients would be required for the training study. Data of patients who participated in the pilot study will be used in the training study. The training study will be carried out in all 12 hospitals.

Validation study Directly after finishing the training study, the validation study will be started in 'new' patients that have not participated in the training study.

Every patient with a suspected thyroid nodule, indicated for additional diagnostic procedures including an ultrasound of the thyroid gland (resulting in the TIRADS classification) followed by a fine-needle aspiration for cytology (resulting in the Bethesda classification), will be asked to participate. We will provide information about the study and obtain a signed informed consent. We expect that in particular, the FNAC might influence the patterns of the VOCs in the exhaled breath, measured by the Aeonose™. For this reason, we will include patients in this study before FNAC will take place.

Patients in the validation study will be asked to participate only once by breathing in the Aeonose™ for five minutes, followed by completing a short questionnaire of known factors that can influence the breathing patterns.

A minimum of 500 patients will be necessary to validate the sensitivity of the pilot study.

This study has no specific benefits for the participating patients. The risks of using the Aeonose are very small. Possible side effects during measurements are dizziness and nausea, usually due to hyperventilation. Other side effects are hypo- or hyper salivation during measurements. Blood will be collected during regular pre-operative blood collection, resulting in no extra skin puncture. Furthermore two quick to answer questionnaires as well as a short case report form (CRF) will be filled in by the participating patients. Using the Aeonose as a non-invasive, rapid and inexpensive diagnostic tool could be a major benefit for patients with thyroid nodules due to the faster and less invasive diagnostic process. Benefits for patients with benign thyroid diseases include the possibility to resign from unnecessary invasive treatments such as (diagnostic) surgery.

We hypothesize that the high negative predictive value of the pilot study will be confirmed in the validation study and expect that implementation of the Aeonose™ in clinical practice will subsequently reduce the number of unnecessary surgeries below 10% for patients with Bethesda ≥ III nodules. For the pilot study on the follow-up, we hypothesize that the Aeonose™ can play an important role in non-invasive detection of recurrent disease. Within several years, analysis of exhaled breath using the Aeonose™ will play an important role in the detection of thyroid cancer and/or its recurrence and will, therefore, have a position in regular clinical decision making

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule requiring additional diagnostic follow-up (TI-RADS/Bethesda)
* Patients with thyroid problems requiring surgery (e.g. goiter)
* AeonoseTM measurement before undergoing cytological puncture or at least 3 days after cytological puncture pre-operatively.
* > 18 year.
* Signed informed consent

Exclusion Criteria:

* Other underlying malignancy, (less than 5 years ago), basal cell carcinoma not included - Unable to participate due to comorbidities (e.g. COPD)
* Not able to understand the information

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who have a scheduled visit in the outpatient clinic of the departments of endocrinology or endocrine surgery for an thyroid nodule needing further diagnostic follow- up will be asked to participate in this study. Patients will be recruited among those visiting the outpatient clinic of the participating hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 4 months
Specificity | 4 months
Positive Predictive Value | 4 months
Negative Predictive Value | 4 months
Area Under the Curve of the Receiver Operating Characteristics Curve | 4 months

SECONDARY OUTCOMES:
Quality of Life | 4 months
  EQ-5D-5L
Burden Thermometer/Problem List | 4 months
  Emotional Burden
Surgical Complications | 4-6 months
  Clavien Dindo Classification
Number of unnecessary surgeries | 4 years
Ease of use of electronic nose | 4 months
  VAS
Sensitivity and Specificity of Molecular Diagnostics | 1 year
  olecular diagnostics on the cytology of thyroid punctures, blood after regular blood sampling, and histology will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, Prof,MD,PhD, Principal Investigator — Maastricht University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the following end products available for further research and verification:
  * Raw data
  * (Several versions of) processed data
  * Data documentation
  * Documentation of the research process, including documentation of all participants
  * Syntaxes
  All data and samples will be stored for 15 years in order to be used for further research in the field of thyroid cancer.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once the associated article is published and/or the project has ended, (part of) the data will be accessible for further research and verification. A possible embargo period is yet to be defined in conjunction with the research team and the eNose company.
Access Criteria: Once the project has ended, the data collection will be publicly accessible without any restrictions.

REFERENCES:
- [Background] Pellegriti G, Frasca F, Regalbuto C, Squatrito S, Vigneri R. Worldwide increasing incidence of thyroid cancer: update on epidemiology and risk factors. J Cancer Epidemiol. 2013;2013:965212. doi: 10.1155/2013/965212. Epub 2013 May 7. PMID 23737785
- [Background] Tessler FN, Middleton WD, Grant EG. Thyroid Imaging Reporting and Data System (TI-RADS): A User's Guide. Radiology. 2018 Apr;287(1):29-36. doi: 10.1148/radiol.2017171240. PMID 29558300
- [Background] Tamhane S, Gharib H. Thyroid nodule update on diagnosis and management. Clin Diabetes Endocrinol. 2016 Oct 3;2:17. doi: 10.1186/s40842-016-0035-7. eCollection 2016. PMID 28702251
- [Background] Cibas ES, Ali SZ; NCI Thyroid FNA State of the Science Conference. The Bethesda System For Reporting Thyroid Cytopathology. Am J Clin Pathol. 2009 Nov;132(5):658-65. doi: 10.1309/AJCPPHLWMI3JV4LA. PMID 19846805
- [Background] Haick H, Broza YY, Mochalski P, Ruzsanyi V, Amann A. Assessment, origin, and implementation of breath volatile cancer markers. Chem Soc Rev. 2014 Mar 7;43(5):1423-49. doi: 10.1039/c3cs60329f. Epub 2013 Dec 4. PMID 24305596
- [Background] de Lacy Costello B, Amann A, Al-Kateb H, Flynn C, Filipiak W, Khalid T, Osborne D, Ratcliffe NM. A review of the volatiles from the healthy human body. J Breath Res. 2014 Mar;8(1):014001. doi: 10.1088/1752-7155/8/1/014001. Epub 2014 Jan 13. PMID 24421258
- [Background] Guo L, Wang C, Chi C, Wang X, Liu S, Zhao W, Ke C, Xu G, Li E. Exhaled breath volatile biomarker analysis for thyroid cancer. Transl Res. 2015 Aug;166(2):188-95. doi: 10.1016/j.trsl.2015.01.005. Epub 2015 Jan 20. PMID 25666355
- [Background] Hoftijzer HC, Heemstra KA, Corssmit EP, van der Klaauw AA, Romijn JA, Smit JW. Quality of life in cured patients with differentiated thyroid carcinoma. J Clin Endocrinol Metab. 2008 Jan;93(1):200-3. doi: 10.1210/jc.2007-1203. Epub 2007 Oct 23. PMID 17956954
- [Background] Barbus E, Pestean C, Larg MI, Piciu D. Quality of life in thyroid cancer patients: a literature review. Clujul Med. 2017;90(2):147-153. doi: 10.15386/cjmed-703. Epub 2017 Apr 25. PMID 28559697
- [Derived] Al-Difaie ZJJ, Scheepers MHMC, Engelen SME, Lubbers T, Havekes B, Bouvy ND. Volatile organic compounds in exhaled breath, blood, and urine detected in patients with thyroid carcinoma using gas chromatography-ion mobility spectrometry-a pilot study. J Breath Res. 2024 Nov 26;19(1). doi: 10.1088/1752-7163/ad89ef. PMID 39437815